CLINICAL TRIAL: NCT02064491
Title: Erlotinib Treatment Beyond Progression in EGFR Mutant or Patients Who Have Responded EGFR TKI in Stage IIIB/IV NSCLC
Brief Title: Erlotinib Treatment Beyond Progression in EGFR Mutant NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Finnish Lung Cancer Group (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETAP; 2013-002049-13 (EudraCT Number)
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; EGFR mutant; Erlotinib; Treatment Beyond Progression
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Drug Therapy; Cisplatin; Carboplatin; Docetaxel; Paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erlotinib and Chemotherapy (Experimental): Intercalated erlotinib in combination with chemotherapy for four to six cycles followed by continuous erlotinib maintenance
  Interventions: Drug: Erlotinib; Drug: Chemotherapy
- Chemotherapy (Active Comparator): Chemotherapy for four to six cycles
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Erlotinib
  Other Names: Tarceva
  Arms: Erlotinib and Chemotherapy
Drug: Chemotherapy
  Other Names: Cisplatin, Carboplatin, Docetaxel, Paclitaxel, Pemetrexed

SUMMARY:
The purpose of this study is to determine whether continuing erlotinib beyond disease progression in combination with chemotherapy is beneficial for NSCLC patients who have EGFR mutant disease or who have responded to EGFR TKI.

DETAILED DESCRIPTION:
A Phase II randomised, multicenter study to assess the efficacy and safety of continuing erlotinib in addition to chemotherapy versus chemotherapy alone in patients who have EGFR mutant or EGFR TKI responsive NSCLC and have progressed on EGFR TKI.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IIIB/IV NSCLC.
* Investigator confirmed progression according RECIST 1.1 during EGFR TKI treatment within 28 days of the randomization
* Activating mutation (G719A/C/S; Exon 19 insertion/deletion; L858R; L861Q) in the EGFR gene or have had at least partial response with EGFR TKI lasting ≥ 6 months
* Performance status: WHO 0-2
* Measurable disease according to RECIST 1.1
* Patients must be able to comply with study treatments
* Women with child-bearing potential and men with reproductive potential must be willing to practice acceptable methods of birth control during the study
* Neutrophils ≥ 1'000/μl, Platelets ≥ 100'000/μl, Alanine amino transferase ≤ 2.5 × Upper limit of normal (ULN) (< 5 × ULN if liver metastases), Alkaline phosphatase ≤ 2.5 × ULN (< 5 × ULN if liver metastases), Serum bilirubin ≤ 1.5 × ULN, Serum Creatinine ≤ 1.5 × ULN.
* Patient must be able to comply with the protocol

Exclusion Criteria:

* RECIST 1.1 defined disease progression for more than 28 days while on previous EGFR TKI treatment.
* Patient has been treated with any investigational agent for any indication within 4 weeks of study treatment.
* Patient has history of hypersensitivity or intolerance to erlotinib or gefitinib.
* Patient has history of hypersensitivity or intolerance to chemotherapeutic agents used in the study.
* Patient with symptomatic central nervous system metastases
* Patient has known active hepatitis B or C, or HIV infection
* Pregnant or breastfeeding.
* Patient with uncontrolled undercurrent illness or circumstances that could limit compliance with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival of the whole study population and in the strata 1-2 | An expected average of 36 weeks after last subject enrolled into our study

SECONDARY OUTCOMES:
Overall Survival | An expected average of 52 weeks after last subject enrolled into our study
Overall Response Rate | An expected average of 36 weeks after last subject enrolled into our study
Rate of non-progression at 9 and 18 weeks | 18 weeks after date of randomization of a last patient
Safety and toxicity | An expected average of 52 weeks after last subject enrolled into our study
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Locations (7):
- Finland (7):
  - Helsinki University Hospital, Espoo
  - Helsinki University Hospital, Helsinki
  - Oulu University Hospital, Oulu
  - Pori Central Hospital, Pori
  - Tampere University Hospital, Tampere
  - Turku University Hopital, Turku
  - Vaasa Central Hospital, Vaasa